CLINICAL TRIAL: NCT00197418
Title: Dual Therapy With High-Dose of Rabeprazole and Amoxicilline Versus Triple Therapy With Rabeprazole, Amoxicilline and Metronidazole as the Second Line Therapy for the Cure of H. Pylori Infection
Brief Title: Second Line Therapy for the Cure of Helicobacter Pylori (H. Pylori) Infection
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamamatsu University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HighdosePPI
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2006-03-21 (Estimated); Status verified 2003-03

CONDITIONS: Helicobacter Infections; Gastritis; Gastric Ulcer; Duodenal Ulcer
Keywords: H. pylori infection
MeSH Terms: conditions — Helicobacter Infections; Gastritis; Stomach Ulcer; Duodenal Ulcer | interventions — Rabeprazole; Amoxicillin; Clarithromycin; Metronidazole

INTERVENTIONS:
Drug: rabeprazole, amoxicillin, clarithromycin, metronidazole

SUMMARY:
Proton pump inhibitors (PPIs) are mainly metabolized in the liver by CYP2C19, one of the cytochrome P450 isoenzymes, which shows a genetic polymorphism associated with enzyme activities. The most essential role of a PPI in H. pylori eradication therapy is to make antibiotics more stable and bioavailable in the stomach by raising intragastric pH to neutral levels.

Most patients who have failed in the eradication of H. pylori infection by triple therapy with a PPI, amoxicillin (AMPC) and clarithromycin (CAM) at standard doses have extensive metabolizer (EM) genotypes of CYP2C19 and/or are infected with CAM-resistant strains of H. pylori.

Four-times daily dosing of a PPI could achieve complete gastric acid inhibition. Dual therapy with 4-times daily dosing of a PPI and AMPC could yield sufficient re-eradication rates in patients with EM genotype of CYP2C19.

Metronidazole (MNZ)-based re-eradication therapy, such as triple PPI/AMPC/MNZ therapy, also achieved high eradication rates and has been recommended as the second line therapy in Japan. But carcinogenic actions of MNZ have been unclear.

The purpose of this study is to compare the re-eradication rates of H. pylori infection by the dual high-dose PPI/AMPC therapy and triple PPI/AMPC/MNZ therapy, and to validate the efficacies of these re-eradication regimens as second line eradication therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with H. pylori infection

Exclusion Criteria:

* Patients without H. pylori infection

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-08

PRIMARY OUTCOMES:
Which treatment yields the higher re-eradication rate of H. pylori infection

SECONDARY OUTCOMES:
Side effects

CONTACTS AND LOCATIONS:
Overall Officials: Naohito Shirai, MD., PhD, Study Chair — Hamamatsu University
Locations (1):
- Hamamatsu University School of Medicine, Hamamatsu, Shizuoka, Japan